CLINICAL TRIAL: NCT05245968
Title: A Phase 1 Study of TAS-116 (Pimitespib) in Combination With Imatinib in Patients With Advanced Gastrointestinal Stromal Tumor
Brief Title: A Study of Pimitespib in Combination With Imatinib in Patients With GIST (CHAPTER-GIST-101)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10058060
Record Dates: First submitted 2022-01-17; First posted 2022-02-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — TAS-116; Imatinib Mesylate; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Part (Experimental): Pimitespib in combination with imatinib
  Interventions: Drug: Pimitespib; Drug: Imatinib
- Expansion Part-A (Experimental): Pimitespib in combination with imatinib
  Interventions: Drug: Pimitespib; Drug: Imatinib
- Expansion Part-B (Experimental): Pimitespib followed by imatinib
  Interventions: Drug: Pimitespib; Drug: Imatinib
- Expansion Part-C (Experimental): Sunitinib
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Pimitespib — Pimitespib will be administered orally in 5 consecutive days followed by 2 days off treatment (QD 5) on an empty stomach at least 1 hour before or 2 hours after a meal. The doses in the Dose Escalation Part will be 80, 120 (starting dose), and 160 mg. The doses used in Arm A will be MTD or recommended dose (RD) based on the information, including the safety and the pharmacokinetics (PK) data in the Dose Escalation Part. In Expansion Part-B, pimitespib will be administered with the starting dose of 160 mg daily.
  Other Names: TAS-116
  Arms: Dose Escalation Part; Expansion Part-A; Expansion Part-B
Drug: Imatinib — Imatinib will be administered orally, after a meal and large glass of water QD. The doses in Dose Escalation Part will be 400 mg or 300 mg (De-escalation). The doses used in Expansion Part-A will be MTD or RD based on information, including the safety and PK data in the Dose Escalation Part. In Expansion Part-B, imatinib will be administered post after pimitespib discontinuation with the starting dose of 400 mg daily.
  Arms: Dose Escalation Part; Expansion Part-A; Expansion Part-B
Drug: Sunitinib — Sunitinib will be administered orally QD with a starting dose of 50 mg, on a schedule of 4 weeks on treatment followed by 2 weeks off, and will be taken with or without a meal in Expansion Part-C.
  Arms: Expansion Part-C

SUMMARY:
This study consists of Dose escalation part and Expansion part. In Dose Escalation Part, the maximum tolerated dose of combination of pimitespib and imatinib in patients with gastrointestinal stromal tumors (GIST) who are judged to be refractory to imatinib, estimate the recommended dose, evaluate safety and pharmacokinetics, and observe the antitumor effect. Expansion part consists of 3 arms. In Arm A, the efficacy and safety will be evaluated, which of the combination of pimitespib and imatinib in patients with GIST who have failed imatinib at doses below the MTD determined in Dose Escalation Part. In Arm B, the efficacy and safety of pimitespib monotherapy will be evaluated and the therapeutic effect of imatinib administration after pimitespib will be evaluated in an exploratory manner. In Arm C, the efficacy and safety of sunitinib monotherapy will be evaluated as reference data.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent
* Histologically confirmed GIST
* Has radiographic progression based on RECIST 1.1 during or within 6 months of the last imatinib administration at enrollment. If surgery/radiotherapy has been performed, radiographic progression based on RECIST 1.1 with imatinib must have been observed after the last surgery /radiotherapy
* Has at least one measurable lesion based on the RECIST version 1.1, except lymph nodes (not dependent on size), which should be chosen as nontarget lesions;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1

Exclusion Criteria:

* Corrected visual acuity < 0.5 (using the International Visual Acuity Measurement Standard) for both eyes
* Received treatment with any other line of therapy besides imatinib for advanced GIST
* History of total gastrectomy and/or whole resection of the small intestine
* A serious illness or medical condition
* Previous or concurrent cancer that is distinct in primary disease or histology from cancer that is being evaluated in this study. However, any previous cancer curatively treated > 5 years before the enrollment can be eligible
* Pregnancy or lactation (including lactation interruption)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) of pimitespib in combination with imatinib | At the end of Cycle 1 (each cycle is 28 days)
Maximum tolerable dose (MTD) of pimitespib in combination with imatinib | At the end of Cycle 1 (each cycle is 28 days)
Progression-free survival (PFS) | approximately 2 years

SECONDARY OUTCOMES:
Overall survival (OS) | approximately 2 years
Overall response rate (ORR) | approximately 2 years
Disease control rate (DCR) | approximately 2 years
Duration of response (DoR) | approximately 2 years
Adverse event (AE) | approximately 2 years
Adverse drug reaction (ADR) | approximately 2 years
Maximum plasma concentration (Cmax) | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
Time to reach maximum plasma concentration (Tmax) | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
Under the plasma concentration-time curve up to the last observable concentration (AUC0-last) | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
λz | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
Half-life (T1/2) | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
Oral clearance (CL/F) | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
Apparent volume of distribution (Vz/F) | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
Mean residence time (MRT) | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
Accumulation ratio | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)
Metabolite ratio | Multiple time points on Day 1 and Day5 or Day12 of Cycle 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (14):
- Australia (2):
  - Flinders Medical Center, Adelaide
  - Alfred Health, Melbourne
- China (2):
  - Beijing Cancer Hospital, Beijing
  - Fudan University, Shanghai Cancer Center, Shanghai
- Japan (6):
  - National Cancer Center Hospital East, Chiba
  - Hokkaido University Hospital, Hokkaido
  - Kumamoto University Hospital, Kumamoto
  - Osaka University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- National University Cancer Institute, Singapore, Singapore
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Linkou Chang Gung Memorial Hospital, Linkou District
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Taiho provides a platform for accepting researchers' requests for sharing anonymized, patient-level, analyzable datasets from articles published in peer-reviewed journals about the primary results from Taiho-sponsored interventional clinical trials in patients in which the medicine and the indication has received marketing approval from regulatory authorities in the United States, the European Union, and/or Japan on or after January 15, 2018.
Supporting Information: Study Protocol, SAP
Time Frame: https://www.taiho.co.jp/en/science/policy/clinical_trial_information_disclosure_policy/index.html
Access Criteria: Access to the clinical trial data is contingent upon approval of a proposed study protocol by an independent review panel and the execution of a data-sharing agreement with the researcher.
URL: https://vivli.org/